CLINICAL TRIAL: NCT01186536
Title: Whey Protein Supp. w/ Resistance Training; Effects on Body Comp. of Young Adults.
Brief Title: Whey Protein, Resistance Training, and Changes in Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Principal Investigator, Richard Washburn, Associate Professor, University of Kansas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSCL16583; DMI01425 (Other Grant/Funding Number: Dairy Management Inc.)
Record Dates: First submitted 2010-03-26; First posted 2010-08-23 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
Keywords: Whey Protein; Soy Protein; Resistance training; Weight Management
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Whey protein supplementation (Experimental): Daily whey protein supplementation
  Interventions: Dietary Supplement: Whey Protein supplement
- Soy Protein supplementation (Experimental): Daily soy protein supplementation
  Interventions: Dietary Supplement: Soy Protein Supplement
- Placebo (Experimental): Daily carbohydrate placebo supplementation
  Interventions: Dietary Supplement: Carbohydrate supplement

INTERVENTIONS:
Dietary Supplement: Whey Protein supplement — 40 g/day of whey protein will be consumed in 2 doses for 9 months (Study duration)
  Arms: Whey protein supplementation
Dietary Supplement: Soy Protein Supplement — 40 g/day of soy protein will be consumed in 2 doses for 9 months (Study duration)
  Arms: Soy Protein supplementation
Dietary Supplement: Carbohydrate supplement — 40 g/day of maltodextrin will be consumed in 2 doses for 9 months (Study duration)
  Arms: Placebo

SUMMARY:
The objective of this project is to determine the effect of 9 months of progressive resistance training with daily whey protein supplements on the body composition (changes in muscle and fat) in young adults. The investigators hypothesize that those individuals who receive whey protein supplements will have larger gains in muscle and larger losses of fat tissue in response to resistance training compared to those who receive supplements of soy or carbohydrate.

DETAILED DESCRIPTION:
Healthy men and women will be recruited to participate in 9 months of supervised resistance training (3 days/wk) and will be randomized to one of three daily supplement groups: Whey protein, soy protein, or carbohydrate control. Body weight, muscular strength and endurance, and resting blood pressure will be assessed at baseline, 3, 6 and 9 months. Body composition will be assessed at baseline, 3, 5, 7, and 9 months. A sub-sample (N = 17 per group, assessed at baseline and 9 months) will be randomly selected for muscle samples of the upper leg to determine changes in the size of muscle fibers, and chemical factors associated with muscle growth. Blood samples will be obtained from sub-sample participants to assess changes in glucose and fat metabolism, as well as other chemicals likely to promote or inhibit muscle growth. We will also assess changes in daily energy expenditure and the use of fuel to produce energy (carbohydrate, fat, protein) that may result from the intervention. We hypothesize that those individuals who receive whey protein supplements will have larger gains in muscle and larger losses of fat tissue in response to resistance training compared to those who receive supplements of soy or carbohydrate.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-39.9
* must be 18- 30 years old
* sedentary
* no medications
* stable weight for at least 3 months

Exclusion Criteria:

* Tobacco/Drug user
* metabolism altering medication
* gain/lost 10lbs in the last 3 months
* current exerciser

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2007-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Body Composition | 9 months
  Changes in body composition will be evaluated by measuring the change in percent body fat, total fat mass, and total lean mass by DEXA.

SECONDARY OUTCOMES:
24 hour energy expenditure and substrate oxidation | 9 months
  24hr energy expenditure and substrate oxidation will be measured by whole room indirect calorimetry
Muscular strength and endurance | 9 months
  One rep max strength will be measured on the chest and leg press.
Resting Metabolic Rate | 9 months
  Resting metabolic rate as measured by indirect calorimetry as kcal/day will be evaluated. Also, substrate oxidation (fat and carbohydrate oxidation) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Washburn, Ph.D., Principal Investigator — University of Kansas
Locations (1):
- Energy Balance Lab, The University of Kansas, Lawrence, Kansas, United States